CLINICAL TRIAL: NCT01395862
Title: Special Drug Use Investigation for ADOAIR (Fluticasone/Salmeterol)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112278
Record Dates: First submitted 2011-07-14; First posted 2011-07-18 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Respiratory Disorders
MeSH Terms: conditions — Respiration Disorders | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients prescribed fluticasone and salmeterol: Patients with asthma prescribed fluticasone and salmeterol for long-term use during study period
  Interventions: Drug: Salmeterol and Fluticasone

INTERVENTIONS:
Drug: Salmeterol and Fluticasone

SUMMARY:
The purpose of this study is to detect adverse drug reactions for long-term use (particularly clinically significant adverse drug reactions) occurring in clinical settings, to examine factors likely to affect the safety and efficacy in the Japanese asthma patients who are treated with fluticasone propionate/salmeterol xinafoate.

ELIGIBILITY:
Inclusion Criteria:

* Must use fluticasone and salmeterol for the first time
* Must use fluticasone and salmeterol for long-term

Exclusion Criteria:

* Patients with hypersensitivity to salmeterol and fluticasone
* Patients with infection which salmeterol and fluticasone is not effective
* Patients with deep mycosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Japanese patients with asthma who are expected to use fluticasone and salmeterol for long-term.
Sampling Method: Probability Sample
Enrollment: 1001 (Actual)
Dates: Start 2007-11; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The number of incidence of adverse events in Japanese asthma patients treated with fluticasone and salmeterol for long-term | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline